CLINICAL TRIAL: NCT00974922
Title: Vitamin D Deficiency, Renin Inhibitor Response, and Vitamin D Supplementation in Patients With Hypertension
Brief Title: Vitamin D Deficiency in Patients With Hypertension
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Administrative/Sponsor Business Decision - terminated - study was not completed
Sponsor: UConn Health (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, William B. White, Professor of Medicine, UConn Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09-166-1; 20090713 (Other: UConn Health Center)
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Results first posted 2018-03-09 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-02

CONDITIONS: Vitamin D Deficiency; Hypertension
Keywords: Vitamin D; Hypertension
MeSH Terms: conditions — Vitamin D Deficiency; Hypertension | interventions — aliskiren; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Phase I: Aliskiren (Active Comparator): Two weeks of single-blind placebo, followed by randomization in a double-blind fashion to Aliskiren 150 mg to 300 mg once daily for 6 weeks
  Interventions: Drug: Aliskiren; Dietary Supplement: Placebo
- Phase I: Cholecalciferol (Active Comparator): Two weeks of single-blind placebo, followed by randomization in a double-blind fashion to Cholecalciferol (3000 I.U.) once daily for 6 weeks
  Interventions: Dietary Supplement: Cholecalciferol; Dietary Supplement: Placebo
- Phase II: Aliskiren and Vitamin D3 (Active Comparator): Aliskiren 150-300 mg orally once daily and Cholecalciferol 3000 I.U. in combination once daily for 6 weeks
  Interventions: Drug: Aliskiren; Dietary Supplement: Cholecalciferol

INTERVENTIONS:
Drug: Aliskiren — 150 mg once daily for 2 weeks, then titrated to 300 mg once daily for 4 weeks
  Other Names: Tekturna
  Arms: Phase I: Aliskiren; Phase II: Aliskiren and Vitamin D3
Dietary Supplement: Cholecalciferol — 3000 I.U. once daily for 6 weeks
  Other Names: Vitamin D3
  Arms: Phase I: Cholecalciferol; Phase II: Aliskiren and Vitamin D3
Dietary Supplement: Placebo — Placebo for two weeks
  Arms: Phase I: Aliskiren; Phase I: Cholecalciferol

SUMMARY:
This study will evaluate the effects of Vitamin D replacement and the effects of an approved medication for hypertension, aliskiren (Tekturna), in patients with high blood pressure who have low levels of vitamin D in their blood. The study will compare the effects of vitamin D or aliskiren alone and in combination on 24-hour blood pressure and biochemical parameters.

DETAILED DESCRIPTION:
This study will assess whether aliskiren will lower clinic blood pressure and 24-hour blood pressure in patients with hypertension and vitamin D deficiency. Additionally, this study will further explore the potential additional effects of adding vitamin D to aliskiren in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Men or women over 21 years of age with a history of Stage 1 or 2 hypertension (defined as a seated diastolic BP ≥ 90 mmHg and < 110 mmHg in the untreated state).
* Patients under treatment for hypertension must be willing and able to discontinue any previous antihypertensive medications for the duration of the study.
* 25-hydroxyvitamin D levels < 30 ng/ml and > 12 ng/ml.
* Women of childbearing potential must be using a medically acceptable form of birth control for the duration of the trial, must have a negative serum pregnancy test at screening, and must have a negative urine pregnancy test within 7 days before initiating aliskiren therapy.

Exclusion Criteria:

* Vitamin D levels < 12 ng/ml
* Known hypersensitivity or allergy to aliskiren
* Clinic blood pressure > 180/110 mmHg
* Known forms of secondary hypertension
* Chronic atrial fibrillation
* Uncontrolled or unstable cardiovascular diseases
* Shift or night workers
* Mid-arm circumference > 42 cm in diameter
* Current or recent (<1 year) alcohol or drug abuse
* Pregnant or lactating women

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William B White, M.D., Principal Investigator — Pat and Jim Calhoun Cardiology Center, University of Connecticut Health Center
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study initiated in 2010, study terminated prematurely by the sponsor in December 2011.
Groups:
- Aliskiren and Vitamin D3 AND Aliskiren Versus Vitamin D3: Study stopped prematurely. Intervention groups combined because data were never unblinded.
Period: Overall Study
Arm/Group | Aliskiren and Vitamin D3 AND Aliskiren Versus Vitamin D3
Started (Group assignment was never unblinded due to discontinuation of study; randomization info unavailable) | 40
Completed | 16
Not Completed | 24
Not completed — study terminated | 24

BASELINE CHARACTERISTICS:
Population: Group assignment was blinded to the PI and was never unblinded due to the discontinuation of the study by the sponsor. Therefore we are unable to determine the number of participants in each group. No data analyses occurred due to lack of any scientific utility of the information.
Groups:
- Aliskiren Versus Vitamin D3 AND Aliskiren and Vitamin D3: Two weeks of single-blind placebo, followed by randomized in a double-blind fashion to aliskiren 150 mg to 300 mg or Vitamin D3 (3000 I.U.) once daily for 6 weeks.
  Aliskiren 150-300 mg orally once daily and Vitamin D3 3000 IU in combination once daily for 6 weeks.
Arm/Group | Aliskiren Versus Vitamin D3 AND Aliskiren and Vitamin D3
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants] — Data not analyzed by groups as group assignment was blinded (and never un-blinded due to discontinuation by the sponsor). There were 30 participants between 18 and 65 years, and 10 participants over 65 years.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 36
    >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.85 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Data not analyzed by groups as group assignment was blinded (and never un-blinded due to discontinuation by the sponsor). There were 25 females and 15 males in total randomized to the study.
  Participants
    Female | 25
    Male | 15

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Ambulatory Diastolic Blood Pressure
Description: The primary endpoint was changes from baseline in 24-hour mean diastolic BP on aliskiren versus vitamin D3 in hypertensive patients with vitamin D deficiency.
Time Frame: six weeks
Population: Study was never completed due to early termination of the trial by sponsor. Data were never analyzed because group assignment was never un-blinded and data lacked any scientific utility.
Groups:
- Aliskiren Versus Vitamin D3 AND Aliskiren and Vitamin D3: Phase I: Two weeks of single-blind placebo, followed by randomization in a double-blind fashion to aliskiren 150 mg to 300 mg or Vitamin D3 (3000 I.U.) once daily for 6 weeks.
  Phase II: Aliskiren 150-300 mg orally once daily and Vitamin D3 3000 IU in combination once daily for 6 weeks.
Arm/Group | Aliskiren Versus Vitamin D3 AND Aliskiren and Vitamin D3
Number analyzed (Participants) | 0

2. Secondary Outcome: Change From Baseline Blood Pressure Measurement in 24-hour Systolic BP, Changes in Awake and Sleep Systolic and Diastolic BP, and Changes From Baseline in Clinic Systolic and Diastolic BP.
Time Frame: 6 weeks
Population: as for outcome 1
Arm/Group | Aliskiren Versus Vitamin D3 AND Aliskiren and Vitamin D3
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the duration of the study ~ 2 years, 6 months
Description: Data not analyzed by groups as group assignment was blinded (and never un-blinded due to discontinuation by the sponsor).
Groups:
- Aliskiren Versus Vitamin D3 AND Aliskiren and Vitamin D3: Phase I: Two weeks of single-blind placebo, followed by randomized in a double-blind fashion to aliskiren 150 mg to 300 mg or Vitamin D3 (3000 I.U.) once daily for 6 weeks.
  Phase II: Aliskiren 150-300 mg orally once daily and Vitamin D3 3000 IU in combination once daily for 6 weeks.
Arm/Group | Aliskiren Versus Vitamin D3 AND Aliskiren and Vitamin D3
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

LIMITATIONS AND CAVEATS:
Study was never completed due to early termination of the trial by sponsor. Data were never analyzed because group assignment was never un-blinded and data lacked any scientific utility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No